CLINICAL TRIAL: NCT00083343
Title: A Multicenter, Open, Noncomparative Study to Estimate the Safety, Tolerability, and Efficacy of Caspofungin Acetate in the Treatment of Adults With Invasive Candida Infections (Excluding Patients With Candidemia as the Sole Site of Infection)
Brief Title: Caspofungin for the Treatment of Non-blood Candida Infections (0991-045)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0991-045; Formerly-0404NBCI; MK0991-045; 2004_102
Record Dates: First submitted 2004-05-20; First posted 2004-05-24 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Candidiasis
MeSH Terms: conditions — Candidiasis | interventions — Caspofungin

INTERVENTIONS:
Drug: MK0991, caspofungin acetate/Duration of Treatment: variable

SUMMARY:
Candida is the most common fungal pathogen identified in hospitalized patients. This study will seek to enroll adult patients (18 years of age or older) with invasive Candida infections (involving deep tissues and organs). The study will not enroll patients whose only site of Candida infection was the bloodstream. Patients that fulfill all study entry criteria will receive a single daily dose of caspofungin. Caspofungin, an intravenous echinocandin antifungal agent, is already approved for the treatment of invasive candidiasis. The dosage strength and duration of caspofungin will be individualized for each patient based on disease, severity of disease and extent of infection.

ELIGIBILITY:
Inclusion Criteria:

* All patients must have at least 1 positive culture for Candida species obtained from an otherwise sterile, non-blood body site within 96 hours of the study entry.
* The patient must also have clinical evidence of Candida infection (e.g., oral temperature >100 degrees Fahrenheit, signs of inflammation from infected site, systolic blood pressure <90) within 96 hours of study entry.
* The patient must be at least 18 years old, and if a woman of child bearing potential, must have a negative serum or urine pregnancy test sensitive to 25 IU HCG prior to enrollment.

Exclusion Criteria:

* Patients whose only site of Candida infection was the bloodstream.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2004-05; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Favorable overall response rate

SECONDARY OUTCOMES:
Favorable overall response rate on Day 10 of caspofungin therapy
Occurance of relapse during the 12 week follow-up period following the completion of all antifungal therapy

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

REFERENCES:
- [Background] Petrovic J, Ngai A, Bradshaw S, Williams-Diaz A, Taylor A, Sable C, Vuocolo S, Kartsonis N. Efficacy and safety of caspofungin in solid organ transplant recipients. Transplant Proc. 2007 Dec;39(10):3117-20. doi: 10.1016/j.transproceed.2007.10.003. PMID 18089335
- Available data/document: CSR Synopsis — http://www.merck.com/clinical-trials/policies-perspectives.html